CLINICAL TRIAL: NCT04931693
Title: Evaluation of Ultrasound Guided Modified Pectoral Nerves Blocks in Transvenous Subpectoral Pacemaker Insertion in Children: Randomized Controlled Trial
Brief Title: PECs Block for Pacemaker Insertion in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Elhaddad, lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-316-2020
Record Dates: First submitted 2021-06-05; First posted 2021-06-18 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Complete Heart Block
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: The patient will be randomly assigned to two equal groups. conventional control group(C) (n=20) where20 children will receive IV paracetamol 20 mg / kg . and Pectoral nerves blocks group (P) (n=20) where 20 children will have PECs Block .
Who Masked: Participant, Care Provider
Masking Description: An online randomization program (http://www.randomizer.org) will be used to generate random list and to allocate patients into two study groups: Random allocation numbers will be concealed in opaque closed envelops. The patient and investigator performing the block and assessing study outcomes will all be blinded to the study group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Active Comparator): conventional control group(C) (n=20) where20 children will receive IV paracetamol 20 mg / kg and atracurium top ups at a dose of 0.1mg/kg. every 30 minutes.
  Interventions: Drug: paracetamol
- PECs (Active Comparator): Pectoral nerves blocks group (P) (n=20) where 20 children will have PECs Block and atracurium top ups upon request.
  Interventions: Procedure: modifiedPECs block

INTERVENTIONS:
Drug: paracetamol — iv post operative analgesia
  Other Names: perfalgan
  Arms: control
Procedure: modifiedPECs block — sonar guided pectoral nerve block
  Other Names: PECs 2 block
  Arms: PECs

SUMMARY:
Evaluation of Ultrasound Guided Modified Pectoral Nerves Blocks in Transvenous Subpectoral pacemaker insertion in Children: Randomized Controlled Trial

DETAILED DESCRIPTION:
BACKGROUND Pectoral nerve blocks (PECs) can reduce intraprocedural anesthetic requirements and postoperative pain. Little is known about the utility of PECs in reducing pain and narcotic use after pacemaker (PM)placement in children. OBJECTIVE The purpose of this study was to determine whether PECs can decrease postoperative pain and opioid use after PM placement in children.

METHODS A single-center controlled trial of pediatric patients undergoing transvenous PM placement between 2020 and 2021 will be performed. Demographics, procedural variables, postoperative pain, and postoperative opioid usage will be compared between patients who undergone PECs and those who undergone conventional anesthetic (Control).

ELIGIBILITY:
Inclusion Criteria:

* congenital or post-operative heart block.

Exclusion Criteria:

* ⦁ Redo patient

  * History of allergic reactions to local anesthetics.
  * Bleeding disorders with International Normalization Ratio( INR) > 1.5 and/or platelets < 50 000.
  * Rash or signs of infection at the injection site.
  * Emergency procedure

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Mean Post-operative pain score by The Face, Legs, Activity, Cry, Consolability scale (FLACC) scale. | immediate, 6,12 ,18 and 24 hours after intervention
  pain score

SECONDARY OUTCOMES:
Total consumption of opioids. | immediate, 6,12 ,18 and 24 hours after intervention
  morphine dose

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy Hospital, Cairo, Egypt

REFERENCES:
- [Result] Anderson R, Harukuni I, Sera V. Anesthetic considerations for electrophysiologic procedures. Anesthesiol Clin. 2013 Jun;31(2):479-89. doi: 10.1016/j.anclin.2013.01.005. Epub 2013 Feb 23. PMID 23711654
- [Result] Yang JK, Char DS, Motonaga KS, Navaratnam M, Dubin AM, Trela A, Hanisch DG, McFadyen G, Chubb H, Goodyer WR, Ceresnak SR. Pectoral nerve blocks decrease postoperative pain and opioid use after pacemaker or implantable cardioverter-defibrillator placement in children. Heart Rhythm. 2020 Aug;17(8):1346-1353. doi: 10.1016/j.hrthm.2020.03.009. Epub 2020 Mar 20. PMID 32201270